CLINICAL TRIAL: NCT04997746
Title: Educational Guidelines Aimed at Pre-frail Elderly From a Family Health Unit, Guarulhos/SP - an Intervention Proposal
Brief Title: Educational Guidelines Aimed at Pre-frail Elderly: Intervention Proposal
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Leonardo Paroche de Matos (Other)
Collaborators: Jadhy Aquino Antunes (Unknown); Bianca Prado de Lima Ramos (Unknown); Daniele Fernanda Mantovani (Unknown); Milla de Castro (Unknown); Victória Sanches Pereira Gimenez (Unknown)
Responsible Party: Sponsor-Investigator, Leonardo Paroche de Matos, Advisor, Leonardo Paroche de Matos
Other Study IDs: 20210724
Record Dates: First submitted 2021-07-24; First posted 2021-08-10 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Health Services for the Aged; Geriatrics
Keywords: Elderly health; Patient Care Team; Family health strategy; Primary Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- educational pharmaceutical guidelines: Qualified listening of participants; General pharmaceutical educational guidelines on the use of medicines; Manufacture and supply of medicine organizer boxes.
  Interventions: Behavioral: Multiprofessional educational interventions
- Nursing Educational Guidelines: Nursing educational guidelines; Qualified listening to participants to resolve doubts related to their comorbidities and aging, bringing comfort in relation to their anxieties.
  Nursing interventions will occur through verbal educational guidelines given individually and according to the reality of each participant assessed by the research, based on the nursing diagnoses obtained from the North American Nursing Diagnosis Association - NANDA-I (definitions and classification 2018- 2020) 11th edition.
  Interventions: Behavioral: Multiprofessional educational interventions
- Nutritional Educational Guidelines: Obtaining anthropometric measurements (weight, in kilograms, height (in meters), knee height, arm and calf circumference (in centimeters) to trace the participant's nutritional profile and, subsequently, personalized and appropriate nutritional guidelines will be carried out for each situation The calculation of the Body Mass Index (BMI) must be performed by dividing the weight (W) in kilograms (kg) by the square of the height (H) in meters (m) and indicates the individual's nutritional status. The BMI for the elderly (LIPSCHITZ, 1994 apud TAVARES et al., 2015) determines underweight less than or equal to 22kg / m2, adequate or eutrophic weight between 22 and 27kg / m2 and overweight result greater than or equal to 27kg / m2 .
  Interventions: Behavioral: Multiprofessional educational interventions; Other: Measurement of anthropometric measurements

INTERVENTIONS:
Behavioral: Multiprofessional educational interventions — Preventive educational interventions
Other: Measurement of anthropometric measurements — Measurement of height (in meters), weight (in kilograms), knee height, arm circumference and calf circumference (in centimeters)
  Groups: Nutritional Educational Guidelines

SUMMARY:
INTRODUCTION: aging is the natural process of deterioration of the reserves of biological systems, human beings are inherent to this process. The elderly population in Brazil grows very quickly, this is due to the drop in fertility, mortality and increased life expectancy. OBJECTIVE: to promote the planning of guiding and educational actions based on the qualification of the frailty of the elderly in the Basic Health Unit of the study through the use of the Multidimensional Assessment of the Elderly in Primary Care (AMPI/AB) tool. METHODOLOGY: an experimental, longitudinal, prospective and analytical study aimed at approximately 20 pre-frail elderly people residing in a specific area of a Family Health Unit in the city of Guarulhos/SP. A survey of data referring to the application of AMPI/AB carried out in 2021 and classified as pre-fragile will be carried out, in order to later select them for research. The participant will receive educational guidance on nutrition, use of medications and nursing guidance as identified as needs. Three months after the intervention, AMPI/AB will be applied in order to observe whether the pre-frail elderly remained or changed category after the experimental multidisciplinary educational interventions.

DETAILED DESCRIPTION:
Experimental, longitudinal, prospective and analytical study aimed at pre-frail elderly people living in a specific area of a Family Health Unit in the city of Guarulhos/SP, developed with the aim of qualifying the health care of the elderly population of the territory of the Basic health Unit in 2021, using the Multidimensional Assessment of the Elderly in Primary Care (MAE/PC questionnaire) as the main data collection instrument, associated with the multidisciplinary educational intervention. Initially, a survey of data referring to MAE/PC carried out in 2021 will be carried out during the routine of care by the authors, in order to identify the elderly who were classified as pre-frail. Data referring to healthy and frail elderly people will be used in the research in a descriptive (quantitative) way. Participants will not be identified, data will be displayed in absolute numbers and frequency.

The educational activities will be carried out through home visits and collection of anthropometric measurements, at which time the Informed Consent Form will be offered to authorize participation in the research. The reference participant and/or caregiver will receive all the necessary information to consciously decide whether or not to participate in the aforementioned research and is free to withdraw at any time, which will not harm any of the parties involved. Participants will also receive educational guidance on nutrition, medication use and nursing guidance as identified as needed.

Three months after the intervention, the MAE/PC questionnaire will be reapplied in order to verify if the participant kept or changed his category after receiving the multidisciplinary recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Time and space oriented seniors;
* Previously classified as pre-fragile;
* Good physical condition for taking anthropometric measurements;
* Who voluntarily agreed to participate in the research;

Exclusion Criteria:

* Elderly classified as "healthy";
* Unsatisfactory physical condition that makes it impossible to measure anthropometric measurements;
* Elderly with amputated limbs;
* In palliative care;
* Who refuse to voluntarily participate in the research

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly participants previously classified as pre-frail based on the Multidimensional Assessment of the Elderly instrument
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Correct use of medications | 3 months
  Adequacy of the correct use of medications with the use of the medication box. subjective outcome
Advances in quality of life (subjective) | 3 months
  Offering guidelines on the health of the elderly, providing them with healthier aging and quality of life, covering critical points of the elderly's health and preventing health problems, providing advances in their self-care and giving them more autonomy, solving doubts related to their comorbidities and the aging process, bringing comfort to their anguish, also including the process of death. Subjective outcome
Calculation of Body Mass Index | 3 months
  Elderly people are expected to remain within the anthropometric parameters according to their age group, based on the calculation of BMI in kg / m ^ 2 (obtained by combining weight (in kilograms) and height (in meters)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Matos, Study Director — Guarulhos City Hall
Locations (1):
- Guarulhos City Hall, Guarulhos, São Paulo, Brazil